CLINICAL TRIAL: NCT02415088
Title: Treatment of Postoperative Pain After Shoulder Surgery. Ultrasound-guided Block of the Axillary and Suprascapular Nerves (Selective Shoulder Block) Versus Ultrasound-guided Interscalene Brachial Plexus Block: An Observer-blinded RCT
Brief Title: Ultrasound-guided Selective Shoulder Block Versus Ultrasound-guided Interscalene Brachial Plexus Block, an RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stessel Björn (Other)
Responsible Party: Sponsor-Investigator, Stessel Björn, MD, Jessa Hospital
Organization: Jessa Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15.26/anesth15.01
Record Dates: First submitted 2015-03-08; First posted 2015-04-14 (Estimated); Last update posted 2016-04-05 (Estimated); Status verified 2016-04

CONDITIONS: Pain, Postoperative
Keywords: Nerve block
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Interscalene block (Active Comparator): block of the plexus brachialis in the interscalene region with local anaesthetics
  Interventions: Procedure: Interscalene block
- Selective shoulder block (Active Comparator): selective block of the suprascapular nerve and the axillary nerve with local anaesthetics
  Interventions: Procedure: Selective shoulder block

INTERVENTIONS:
Procedure: Interscalene block — block of the plexus brachialis in the interscalene region with local anaesthetics
  Arms: Interscalene block
Procedure: Selective shoulder block — selective block of the suprascapular nerve and the axillary nerve with local anaesthetics
  Arms: Selective shoulder block

SUMMARY:
This is a randomised, observer-blinded trial to compare selective shoulder block with interscalene block. Both blocks will be placed using an ultra-sound guided technique.

Primary outcome measures will be postoperative pain scores and use of rescue opioids. Secondary outcome measures will be pre- and postoperative occurence of motor deficit of the arm and dyspnea, quality of sleep in the first night after surgery as measured by a numeric rating scale and overall satisfaction with pain therapy as measured by the International Pain Outcomes questionnaire and an NRS-score (0 = not satisfied at all and 10 = very satisfied).

Primary and secondary outcome measures will be assessed during the first 24hours after surgery (assessment in the postanesthetic care unit (PACU) directly after admission and before discharge and in the surgical ward at 4, 8 and 24 hours after surgery).

Overall satisfaction with pain therapy will be assessed 48hours after surgery.

An interscalene block is a block of the plexus brachialis in the interscelene triangle (by injecting a local anesthetic around the nerve plexus).

A selective shoulder block is a block of the suprascapular and axillary nerves (by injecting a local anesthetic around these nerves).

DETAILED DESCRIPTION:
This is a randomised, observer-blinded trial to compare selective shoulder block with interscalene block.

The goal of this study is to compare ultrasound-guided selective shoulder block (regional anesthesia of the suprascapular and axillary nerves) with ultrasound-guided interscalene block after arthroscopic shoulder surgery.

More specific, this study is designed to compare postoperative pain scores, use of opioids, pre- and postoperative occurence of motor deficit of the arm and dyspnea, quality of sleep in the first night after surgery as measured by a numeric rating scale and overall satisfaction as measured by the International Pain Outcomes questionnaire and an NRS-score (0 = not satisfied at all and 10 = very satisfied).

Primary and secondary outcome measures will be assessed during the first 24hours after surgery (assessment in the postanesthetic care unit (PACU) directly after admission and before discharge and in the surgical ward at 4, 8 and 24 hours after surgery).

Overall satisfaction with pain therapy will be assessed 48hours after surgery.

Continuous interscalene brachial plexus block is considered to be the standard treatment for postoperative pain after shoulder surgery. With interscalene block a local anesthetic is injected around the nerve plexus supplying motor and sensory innervation to the upper limb. Disadvantages are an extensive motor and sensory block of the upper limb and paresis of the diaphragm sometimes provoking dyspnea.

Since 2007 newer techniques are described, for example selective block of the suprascapular nerve and the axillary nerve. These two nerves supply most of the shoulder joint with motor and sensory innervation, but have no function in the distal part of the upper limb. The risk of loss of innervation to the diaphragm is avoided with this selective shoulder block. Hence, possible breathing disorders are avoided. Previous studies have concluded that the selective shoulder block is a safe technique and is effective to reduce postoperative pain after arthroscopic shoulder surgery. Moreover, studies also suggest that selective shoulder block has a longer duration, less fluctutations in pain score and less rebound pain after fading of the regional anesthesia.

With this study the investigators want to compare the effect of this newer technique with the single shot interscalene plexus block. Therefore the investigators will allocate the patients to two groups for comparison. One group will receive interscalene plexus block and the other group will receive a selective shoulder block. The used local anesthetic will be the same in both groups, that is ropivacaine 0,75% with a total volume of 20 ml.

Both blocks will be placed using an ultra-sound guided technique. In previous studies a blind technique, based on anatomical reference points or nerve stimulation, has been used to place the selective shoulder block. As both blocks will be placed with an ultrasound-guided technique, the anesthesiologist will have a direct view of the location of the needle. With this technique there is less risk for accidental intravascular injection or nerve injury. Also there is greater probability of success and faster implementation of the block.

Indepent of the technique used, the pain that the patient may experience will be reduced to a minimum. Therefore the patient wlll be supplied with a PCIA system (patient controlled intravenous analgesia), next to the standard pain relievers (paracetamol, anti-inflammatory medication). This PCIA system is a pump system with piritramide (Dipidolor®, an opioid) connected with the infusion line. The system is set up in a way that, within certain limits, the patient can decide for him/herself when pain treatment is provided.

This is a monocentric, prospective, randomised and observer-blinded study. Patients included will be randomised in two groups. One group will receive the ultrasound-guided single shot interscalene block, the other group will receive the ultrasound-guided selective shoulder block (axillary nerve and suprascapular nerve). The patient is not strictly blinded as there are two injections needed for the selective shoulder block, compared to only one injection for the interscalene block. The data collector (per- and postoperative) will be blinded, as he will not be informed about which block is performed. This in order to avoid bias.

ELIGIBILITY:
Inclusion Criteria:

* elective arthroscopic shoulder surgery
* elective hospital admission for one night
* age > 18 years and < 75 years
* American Society of Anesthesiologists (ASA) physical status classification 1, 2 of 3.

Exclusion Criteria:

* pregnancy
* severe obesity ( BMI > 35)
* severe COPD (Gold≥ 3) or restrictive (FEV1 < 50%) lungdisease
* coagulation disorders
* diabetes mellitus
* previous injury or surgery of the involved shoulder
* pre-existing neuropathy or myopathy of the involved arm
* allergy or contra-indication for the medication used in the study
* preoperative use of opioids
* infection at the puncture site
* inability to understand or speak Dutch
* inability to understand the PCIA system
* inability to understand the NRS pain score system
* refusal to participate in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-04; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Pain Score as measured by Numeric Rating Scale | 24hours
Use of piritramide as documented by the PCIA (patient controlled intravenous analgesia) system | 24hours

SECONDARY OUTCOMES:
Subjective feeling of dyspnea as measured by a numeric rating scale | 24hours
Motor deficit after nerve block as measured by Medical Research Council scale | 24hours
Quality of sleep in the first night after surgery as measured by a numeric rating scale | 24hours
Overall satisfaction as measured by the International Pain Outcomes questionnaire | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Schoorens, MD, Principal Investigator — Jessa Hospital
Locations (1):
- Jessaziekenhuis Hasselt, Hasselt, Limburg, Belgium

REFERENCES:
- [Derived] Neuts A, Stessel B, Wouters PF, Dierickx C, Cools W, Ory JP, Dubois J, Jamaer L, Arijs I, Schoorens D. Selective Suprascapular and Axillary Nerve Block Versus Interscalene Plexus Block for Pain Control After Arthroscopic Shoulder Surgery: A Noninferiority Randomized Parallel-Controlled Clinical Trial. Reg Anesth Pain Med. 2018 Oct;43(7):738-744. doi: 10.1097/AAP.0000000000000777. PMID 29659438